CLINICAL TRIAL: NCT02364635
Title: PRC 4016 (Icosabutate) - A Phase I, Single-Blind, Placebo Controlled, Single Oral Dose, Safety, Tolerability and Pharmacokinetic Study in Healthy Subjects
Brief Title: Icosabutate - A Phase I, Single Oral Dose, Safety, Tolerability and Pharmacokinetic Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pronova BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: CTN401614104
Record Dates: First submitted 2015-01-22; First posted 2015-02-18 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Healthy
Keywords: Phase I pharmacokinetics and safety study
MeSH Terms: interventions — icosabutate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Icosabutate dose 1 (Experimental): Dose 1
  Interventions: Drug: icosabutate
- Icosabutate dose 2 (Experimental): Dose 2
  Interventions: Drug: icosabutate
- Icosabutate dose 3 (Experimental): Dose 3
  Interventions: Drug: icosabutate
- Placebo (Placebo Comparator): Placebo (medium chain triglycerides)
  Interventions: Drug: icosabutate
- Icosabutate dose 4 (Experimental): Dose 4
  Interventions: Drug: icosabutate

INTERVENTIONS:
Drug: icosabutate — Single dose at each dose levet
  Other Names: PRC-4016

SUMMARY:
PRC 4016 (Icosabutate) - A Phase I, Single-Blind, Placebo Controlled, Single Oral Dose, Safety, Tolerability and Pharmacokinetic Study in Healthy Subjects

Objective:

* To assess the safety and tolerability of single ascending oral doses of icosabutate in healthy subjects
* To evaluate the pharmacokinetic (PK) parameters of icosabutate in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* males of females
* any ethnic origin
* Age 18-55 years
* BMI 18.0 - 33.0 kg/m2
* generally in good health
* signed informed consent

Exclusion Criteria:

* males or females not willing to use appropriate contraception
* recent blood donation
* recent blood received
* high consumption of alcohol
* high consumption of tobacco
* subjects who have engaged in heavy exercise last two weeks
* prescribed systemic or topical medication taken recently, or supplements/remedies interfering with study procedures or safety
* other medication know to alter drug absorption or elimination
* abnormal heart rate or blood pressure or 12-lead ECG
* significant history of drug allergy, or hypersensitivity to treatment ingredients
* ocular disorder requiring topical ocular therapy, or recent allergic eye disease
* other significant medical history or physical findings

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2015-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic assessments of icosabutate - AUC | 0-36 hour
  Exposure level of icosabutate measured as Area Under the Curve (AUC)
Pharmacokinetic assessments of icosabutate - Cmax | 0-36 hour
  Maximum observed plasma concentration of icosabutate (Cmax)
Number of patients with Adverse Events | During the 36 hour assessment, and at post-study visit day 5-7
  Clinically significant abnormalities found during the course of the study will be followed up until they return to normal or can be clinically explained

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Brooks, MD, Principal Investigator — Covance
Locations (1):
- Covance Clinical Research Unit (CRU) Ltd., Leeds, United Kingdom